CLINICAL TRIAL: NCT07350993
Title: Evaluation of the Effect of Music on the Management of Dental Anxiety in Children: Turkish Validity and Reliability Study of the CEDAM-A Randomized Controlled Clinical Trial
Brief Title: Effect of Music on Dental Anxiety in Children: Turkish Validation of the CEDAM
Acronym: MUSIC-CEDAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şevval Çakıcı (Other)
Responsible Party: Sponsor-Investigator, Şevval Çakıcı, Assistant Professor,DDS, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAKICIAKKOC-DENTALANXIETY; 2024/05-32 (Registry Identifier: Kutahya Health Sciences University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2025-12-17; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Dental Anxiety
Keywords: Behavior guidance; Dental anxiety; Validity; Reliability; Music

STUDY DESIGN:
Intervention Model Description: The study used a parallel-group design with two groups: a music intervention group and a control group. Participants in the intervention group listened to classical instrumental music during dental treatment, while the control group received treatment without music.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention Group (Experimental): Children will listen to classical music during dental treatment to assess the effect on dental anxiety.
  Interventions: Behavioral: Music Listening Intervention
- Control Group (No Intervention): Children will receive dental treatment without any music intervention.

INTERVENTIONS:
Behavioral: Music Listening Intervention — Children will listen to classical instrumental music through headphones during the dental procedure to reduce anxiety levels.
  Other Names: Classical Music Listenin
  Arms: Music Intervention Group

SUMMARY:
The study will consist of two phases. In the first phase, the validity and reliability of the CEDAM scales will be assessed in children aged 9-16 years using item analysis, content and construct validity, internal consistency, and test-retest reliability.

In the second phase, the effect of music will be evaluated in a randomized controlled trial involving children aged 9-12 years. The study will employ a three-session design with progressively increasing procedural invasiveness. In the final session, the control group will receive basic behavior guidance, while the intervention group will additionally listen to music during the dental procedure.

Perioperative anxiety will be assessed using the Children's Anxiety Meter-State (CAM-S), Children's Emotional Manifestation Scale (CEMS), and CEDAM-8. A conceptual model will be used to examine the relationships between music intervention, preoperative anxiety, intraoperative anxiety, and postoperative anxiety.

DETAILED DESCRIPTION:
The study will be conducted in two sequential phases. In the first phase, the cross-cultural validity and reliability of the Children's Experiences of Dental Anxiety Measure (CEDAM) will be assessed in children aged 9-16 years. In the second phase, a subgroup of children aged 9-12 years will be selected from the Phase 1 sample to participate in a randomized controlled trial evaluating the effect of a music intervention on perioperative dental anxiety. Only children requiring at least a second and third dental appointment will be eligible for Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9-16 years
* Systemically healthy children
* Native Turkish speakers
* Written informed consent obtained from both the child and a parent or legal guardian

Exclusion Criteria:

* Presence of any mental or physical disability
* History of psychiatric or developmental disorders
* Known allergies
* Use of medications

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Children's Anxiety Meter-State (CAM-S) Score | Baseline (5 minutes before start of the dental procedure), intra-procedural (immediately after administration of local anesthesia), and post-procedural (5 minutes after completion of the dental procedure)
  Description: A projective measurement tool consisting of a thermometer-like scale with 10 horizontal lines. The scale evaluates state anxiety levels. Scores range from 1 to 10, where higher scores indicate higher levels of anxiety.
  Unit of Measure: CAM-S score
Children's Emotional Manifestation Scale (CEMS) Score | Periprocedural (from seating in the dental chair to completion of the dental procedure)
  Description: An observational behavioral assessment tool that evaluates five main categories: facial expression, vocalization, activity, interaction, and cooperation. Each category is rated on a 5-point scale. Total scores range from 5 to 25, where higher scores indicate higher levels of behavioral anxiety.
  Unit of Measure: CEMS score
Children's Experiences of Dental Anxiety Measure (CEDAM-8) Score | Baseline (5 minutes before start of the dental procedure) and post-procedural (5 minutes after completion of the dental procedure)
  Description: A psychometric tool based on cognitive-behavioral therapy. It consists of 8 questions assessing thoughts, behaviors, physical symptoms, and feelings related to dental anxiety. Responses are recorded on a 3-point Likert scale. Total scores range from 8 to 24, where higher scores indicate greater dental anxiety.
  Unit of Measure: CEDAM-8 score

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Kütahya, Kütahya, Turkey (Türkiye)